CLINICAL TRIAL: NCT06256068
Title: Determinants of Physical Activity Level in Pediatric Oncological Patients Treated With Cardiotoxic Therapy - a Study Protocol
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Julia Haponiuk-Skwarlińska, Principal investigator, Medical University of Warsaw
Other Study IDs: KB/54/A2023
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms
Keywords: exercise capacity; physical activity; cardiotoxicity; childhood cancer; pediatric oncology
MeSH Terms: conditions — Neoplasms; Motor Activity; Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- study group: Study Group: 150 children aged 1 to 5 years, who have completed cancer treatment involving cardiotoxicity risk factors, are now being monitored in follow-up observations.
  The participants' examination will include:
  An exercise capacity test (CPET) to assess exercise capacity
  An extended ALPHA (Assessing Levels of Physical Activity) health-related fitness test battery to evaluate physical function
  Echocardiography to assess cardiac function
  Questionnaires, including the Pediatric Quality of Life Inventory (PedsQL) to measure quality of life, the Physical Activity and Leisure Motivation Scale (PALMS) to assess motivation for physical activity, and an original questionnaire to evaluate lifestyle, socio-demographic factors, self-efficacy, and anthropometric factors
  Use of an ActiGraph GT3X Accelerometer-a wearable device attached to an elastic belt-to monitor physical activity levels for 14 days
- control group: Control Group: 150 children aged 1 to 5 years, who have completed cancer treatment without cardiotoxicity risk factors, are also under follow-up observation. The examination for this group will include:
  An exercise capacity test (CPET) to assess exercise capacity
  An extended ALPHA health-related fitness test battery to evaluate physical function
  Echocardiography to assess cardiac function
  Questionnaires, including the Pediatric Quality of Life Inventory (PedsQL) to measure quality of life, the Physical Activity and Leisure Motivation Scale (PALMS) to assess motivation for physical activity, and an original questionnaire to evaluate lifestyle, socio-demographic factors, self-efficacy, and anthropometric factors
  Use of an ActiGraph GT3X Accelerometer to measure physical activity levels for 14 days.

SUMMARY:
Cancer treatment in children is generally effective, but unfortunately, it often comes with side effects-unwanted negative impacts. Some medications used in cancer treatment, while beneficial in treating the disease, can have harmful effects on the heart and reduce a child's ability to tolerate physical activities such as climbing stairs, walking fast, running, or exercising. Physical activity is crucial for the proper growth and development of children, as well as for their future health as adults. The heart plays a vital role in pumping blood throughout the body, and its proper function is key to a person's ability to engage in physical activity.

The goal of this study is to understand the factors that influence physical activity levels in children who have undergone cancer treatment with methods that may be harmful to the heart. The researchers aim to investigate how these treatments affect the physical activity levels of these children.

The main questions the study seeks to answer are:

Do children who have undergone cancer treatment involving heart-toxic methods show lower levels of daily physical activity compared to children treated with non-toxic methods?

Is the level of physical activity influenced by heart-toxic treatment, or by other factors such as exercise capacity (measured through physical tests like treadmill or standing bike tests), quality of life, lifestyle, social and demographic factors, body type, or knowledge and motivation related to the positive effects of physical activity?

Participants will:

Complete a questionnaire

Perform an exercise test on a treadmill or standing bike to measure exercise capacity

Take part in the ALPHA physical fitness test, which includes simple exercises like jumping and running

Be measured for height and weight

Undergo a hand-grip test using a hand dynamometer

Wear an activity tracker for 14 days

Have an echocardiogram (ultrasound of the heart)

Researchers will compare 150 children treated with heart-toxic methods for cancer to 150 children treated with non-toxic methods. The children will be between 8 and 18 years old and will be 1 to 5 years post-cancer treatment.

The researchers hope that identifying the factors affecting physical activity levels in children treated with heart-toxic methods may improve cancer therapies for children, reduce side effects, and ultimately lead to increased physical activity. This would help promote better growth and overall health for these children in the future.

ELIGIBILITY:
Study group Inclusion criteria

1. age 8-18 years,
2. diagnosis of, and completed treatment for, cancer >1 year and <5 years ago,
3. remission of the cancer,
4. treatment involving use of anthracyclines, kinase inhibitors targeting BRC-ABL, hemopoietic stem cell transplantation, and radiotherapy (TBI or mediastinum irradiation),
5. at least 6 weeks since the last signs or symptoms of an infection,
6. written consent signed by the parents/guardians and by patients aged ≥16 years. Control group

a. the same as for the experimental group and, b. cancer treatment without use of anthracyclines, kinase inhibitors targeting BRC-ABL, hemopoietic stem cell transplantation, and radiotherapy (TBI or mediastinum irradiation).

Both groups Exclusion criteria

1. history of another cancer and its treatment with or without the use of anthracyclines, kinase inhibitors targeting BRC-ABL, hemopoietic stem cell transplantation, and radiotherapy (TBI or mediastinum irradiation),
2. significant physical disability or a muscosceletal disorder at the time of the enrollment (congenital or as a consequence of treatment, especially neurological complications and lower extremities conditions and amputation),
3. excessive malaise (at the time of the enrollment),
4. intellectual disability (on the level that disenables the participant from understanding and cooperation during the CPET procedure or ALPHA test),
5. active acute inflammatory disease including the following: autoimmunological, neurological, pulmonological, endocrinological, cardiovascular, and gastrointestinal,
6. platelet count < 20 G/L,
7. hemoglobin concentration < 9g /dL,
8. severe residual changes (protein loss syndrome, peritoneal, pericardial or pleural effusion, arrhythmia, metabolic disorders),
9. previously diagnosed congenital heart defects or other heart diseases (including cardiomyopathy, heart failure, arrythmia),
10. relapse of the cancer at the time of enrollment to the study,
11. severe malnutrition <3 standard deviation (SD) body mass index (BMI) weight for age,
12. chronic concomitant diseases that could affect the CPET outcome, especially endocrinological, neurological, gastrointestinal, and pulmonological*,
13. lack of patient cooperation.

    * endocrinological - decompensated thyroid disease, decompensated diabetes with hypoglycemia; neurological - conditions disabling the CPET performance due to musculoskeletal system alteration, uncontrolled epilepsy, myopathy; gastrointestinal - marasmus, decompensated hepatic insufficiency; pulmonological - asthma, interstitial lung disease, post-infection bronchiolitis obliterans (PIBO) - additionally, pulmonary embolism, lower extremity phlebitis, kidney failure.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study group will consist of 144 children >1 year and <5 years from a cancer treatment completion involving car-diotoxicity risk factors and are now in the follow-up observation at the outpatient clinic.
  The control group is going to involve 144 children who are >1 year and <5 years from a cancer treatment completion without cardiotoxicity risk factors and are now in the follow-up observation.
  The sample size was calculated for an unmatched case-control study with the input parameters of a 2-sided confidence level of 0.95, power 80%, ratio of controls to cases 1:1, and odds an ratio of 2.0. The sample size calculation by Fleiss with CC method showed 144 participants for each group. Considering a dropout rate of 10%, the total sample size required is 300.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity level measured by the accelerometer | 14 days measurement for 1 individual
  The primary outcome of interest is the PA level measured by the accelerometer and the assessment of the World Health Organization (WHO) pediatric, age-adjusted PA achievement norms.

SECONDARY OUTCOMES:
Percentage of participants disqualified from CPET | Measured at the enrollment
  Percentage of participants disqualified from CPET examination - secondary outcome is the assessment of the proportion of eligible pediatric oncology patients for CPET examination as well as the reasons and characteristics of the patients that were excluded from CPET examination,
Exercise capacity measured in CPET | Measured at the enrollment
  Exercise capacity measured in CPET - maximal/peak oxygen consumption (VO2max/peak) below 47 mL/kg/min for boys and 42 mL/kg/min for girls will be defined as the EC alterations - secondary outcome is the maximal/peak oxygen consumption (VO2max/peak) measurement and defining the EC among the participants,
Physical function in the ALPHA test battery | Measured at the enrollment
  Assessment of the fitness in the extended ALPHA (Assessing Levels of Physical Activity) health-related fitness test battery - defining the fitness level as low, moderate, or high (33, 34) - secondary outcome is the assessment of the physical fitness among the study group in the extended ALPHA test and defining its level,
Cardiac function | Measured at the enrollment
  In cardiological assessment: global longitudinal strain (GLS), global radial strain (GRS), and global circumferential strain (GCS) below average for age, left ventricle diastolic diameter (LVDd) exceeding the normal limit, and ejection fraction (EF) 55% or less will be defined as the lowered systolic function, as well as in the comparison to the control groups - secondary outcome is the contractile function assessment of the heart among the study group and in comparison to the control group.

IPD SHARING:
Plan to Share IPD: No
The raw data (individual participant data (IPD) collected in this study) supporting the conclusions of this article will be made available by the authors, without undue reservation.

REFERENCES:
- [Derived] Haponiuk-Skwarlinska J, Gasior JS, Albrecht K, Laguna P, Werner B. Determinants of physical activity level in pediatric oncological patients treated with cardiotoxic therapy - a study protocol. BMC Pediatr. 2025 May 5;25(1):355. doi: 10.1186/s12887-025-05714-5. PMID 40320516